CLINICAL TRIAL: NCT03022565
Title: Proof of Concept Study of Vorinostat, A Histone Deacetylase Inhibitor, in Patients With Class 2 High Risk Uveal Melanoma
Brief Title: Vorinostat in Patients With Class 2 High Risk Uveal Melanoma
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Investigator Decision
Sponsor: University of Miami (Other)
Collaborators: University of Miami Sylvester Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, J. William Harbour, MD, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20160653
Record Dates: First submitted 2016-12-21; First posted 2017-01-16 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Uveal Melanoma
Keywords: Uveal Melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vorinostat (Experimental): Vorinostat:
  * 400 mg orally, once daily for 15 days.
  Interventions: Drug: Vorinostat

INTERVENTIONS:
Drug: Vorinostat — Study participants who meet the criteria of Class 2 uveal melanoma and no radiologic evidence of metastases will be treated with 400 mg of Vorinostat daily for 15 days.
  Other Names: Zolinza

SUMMARY:
This proof-of-concept study will evaluate the ability of vorinostat to induce the transformation of Class 2 uveal melanoma cells into a cell phenotype that resembles normal melanocytes.

DETAILED DESCRIPTION:
This is a proof of concept, single-center, open-label study of an FDA-approved drug, vorinostat, a Histone deacetylase (HDAC) inhibitor, for patients with Class 2, high-risk uveal melanoma with localized eye tumors. The primary aim is to test if vorinostat can transform aggressive class 2 uveal melanoma cells into cells that look more like normal melanocytes as observed in the laboratory. Uveal melanoma patients that meet the inclusion criteria outlined in this protocol will be consented and asked to provide a fine needle aspiration (FNA) biopsy of their uveal melanoma primary tumor. This biopsy will be submitted for gene expression analysis to determine the phenotype of the tumor. A total of 10 patients who meet the criteria of Class 2 uveal melanoma and no radiologic evidence of metastases will be treated with 400 mg of vorinostat daily for 15 days. On Day 15, patients will be asked to provide a second FNA biopsy prior to receiving the standard of care local definitive therapy either plaque radiotherapy or enucleation.

ELIGIBILITY:
Inclusion Criteria:

1. Uveal melanoma tumor determined by ophthalmic ultrasound or clinical assessment.
2. Class 2 uveal melanoma
3. No evidence of metastatic disease.
4. Age ≥18 years.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
6. Life expectancy of greater than 3 months.
7. Able to swallow and retain orally-administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
8. Patients must have normal organ and marrow function as defined below:

   * Absolute neutrophil count (ANC) >1,500 cells/mm³
   * Platelet count >100,000/mm³
   * Hemoglobin >10.0g/dL
   * Aspartate transaminase (AST) and/or Alanine transaminase (ALT) < 3x upper limited of normal (ULN)
   * Total bilirubin < 2x ULN
   * Hemoglobin A1C ≤ 5.7%
   * Alkaline phosphatase < 3x ULN
   * Serum creatinine < 2x ULN or a creatinine clearance > 60 mL/min
   * Note: Patients with hyperbilirubinemia clinically consistent with an inherited disorder of bilirubin metabolism (e.g., Gilbert syndrome) will be eligible at the discretion of the treating physician and/or the principal investigator.
9. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation until 4 months after completion of study drug administration. Women of child-bearing potential must have a negative serum or urine test at time of enrollment. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study therapy, and 4 months after completion of study drug administration.
10. Willingness to comply with all the visits and procedures (including providing all biological specimens) as required by the protocol and the informed consent form (ICF).
11. Ability to understand the investigational nature, potential risks and benefits of the research study and to provide valid written informed consent.

Exclusion Criteria:

1. Definitive therapy of the primary uveal melanoma by either surgery or radiotherapy
2. History of another malignancy except for those who have been disease-free for 3 years, or patients with a history of completely resected non-melanoma skin cancer and/or patients with indolent secondary malignancies not requiring active therapy, are eligible. Consult the study Principal Investigator if unsure whether second malignancies meet the requirements specified above.
3. Any major surgery or extensive radiotherapy, chemotherapy with delayed toxicity, biologic therapy, or immunotherapy within 21 days prior to initiation of study therapy.
4. History of prior vorinostat use.
5. Use of other investigational drugs within 28 days
6. Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to vorinostat (i.e. HDAC inhibitor hydroxamates such as panobinostat and belinostat).
7. A QT interval corrected (QTc) for heart rate using the Bazett's formula (QTcB) ≥ 480 msec. Concurrent administration of vorinostat and agents that can cause QTc prolongation is not permitted.
8. Concurrent administration of vorinostat and other HDAC inhibitors is not permitted due to the increased risk of thrombocytopenia and gastrointestinal bleeding.
9. Patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with vorinostat.
10. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infections, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with the study requirements.
11. History of pulmonary embolism (PT) or deep-vein thrombosis (DVT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-01-29 (Actual); Study Completion 2020-01-29 (Actual)

PRIMARY OUTCOMES:
Degree of transformation from a class 2 phenotype into a cell phenotype that resembles normal melanocytes. | From Baseline to 15 Days of Protocol Therapy, Up to 4 Weeks
  The investigators will analyze gene expression results from fine needle aspirate biopsies performed at baseline prior to vorinostat therapy and post-treatment (on Day 15, after the planned 15 days of vorinostat therapy).
Proportion of patients whose tumors transformed from a class 2 phenotype into a cell phenotype that resembles normal melanocytes. | From Baseline to 15 Days of Protocol Therapy, Up to 4 Weeks
  Through gene expression analysis, the investigators will determine the proportion of patients whose tumors transformed from a Class 2 phenotype into a cell phenotype that resembles normal melanocytes.

SECONDARY OUTCOMES:
Toxicity During Protocol Therapy | Up to 1 Month Post-Treatment Completion
  Rate of adverse events (AEs) and serious adverse events (SAEs) experienced by study participants during Vorinostat therapy and up to one month after Vorinostat treatment completion.
Tumor size before and after Vorinostat therapy | From Baseline to 15 Days of Protocol Therapy, Up to 4 Weeks
  Tumor size will be determined before and after Vorinostat therapy by B-Scan ultrasonography.
Recurrence-free survival (RFS) | Up to 5 Years Post-Treatment Completion
  Recurrence-Free Survival (RFS) in Study Participants. RFS is defined as the duration of time from start of treatment to time of disease recurrence or death, whichever occurs first.
Overall survival (OS) | Up to 5 Years Post-Treatment Completion
  Overall Survival (OS) in Study Participants. OS is defined as the length of time from date of start of Vorinostat treatment to death.
Disease Specific Survival (DSS) | Up to 5 Years Post-Treatment Completion
  Disease Specific Survival (DSS) in Study Participants. DSS is defined as the time from start of Vorinostat treatment to death due to disease.

OTHER OUTCOMES:
Global histone acetylation levels in peripheral blood mononuclear cells (PBMCs) before and after Vorinostat therapy. | From Baseline to 15 Days of Protocol Therapy, Up to 4 Weeks
  Global histone acetylation levels in peripheral blood mononuclear cells (PBMCs) will be measured at baseline (Day 1, before Vorinostat treatment) and post-treatment (day 15 after completion of Vorinostat therapy).

CONTACTS AND LOCATIONS:
Overall Officials: J. William Harbour, MD, Principal Investigator — University of Miami

IPD SHARING:
Plan to Share IPD: No